CLINICAL TRIAL: NCT05185453
Title: Strengthening Adolescent-Adult Networks to Reduce Youth Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Culyba, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY21030140; 1K23HD098277-01 (NIH)
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-06

CONDITIONS: Violence in Adolescence; Social Interaction; Coping Skills; Adolescent Behavior
Keywords: social networks; social support; violence prevention
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: This pilot community-partnered cluster-randomized trial will examine the feasibility and acceptability of a social network-based youth violence prevention program called Strengthening Connections for Change for youth ages 13-17 and their key adult supports. The study will be located in four lower resource Pittsburgh, Pennsylvania neighborhoods ('clusters') randomized to receive either the Strengthening Connections for Change program (i.e. intervention neighborhoods, n=2) or to a job skills training program (i.e. control neighborhoods, n=2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening Connections for Change (Experimental): Strengthening Connections for Change uses a group discussion format with activities that explore identity, adolescent-adult relationships, social networks, and community engagement. Youth invite their self-identified key adult supports to jointly participate in programming and curriculum includes youth-focused, adult-focused and jointly focused activities designed to build leadership skills, enhance intergenerational networks, challenge attitudes towards violence and retaliation, and reduce violence involvement. Through 12 sessions (2 hours/session) delivered weekly, Strengthening Connections offers leadership development coupled with strengths-based youth violence prevention programming.
  Interventions: Behavioral: Strengthening Connections for Change
- Job Readiness Training (Active Comparator): Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth. Participants receive a 12 session job readiness training with linkages to businesses and employment opportunities. Discussions include a wide range of topics related to career exploration and job readiness.
  Interventions: Behavioral: Job Readiness Training

INTERVENTIONS:
Behavioral: Strengthening Connections for Change — Strengthening Connections for Change is a 12-session curriculum designed to strengthen adolescent-adult support networks, build leadership skills, foster community engagement, and challenge attitudes and behaviors that foster violence involvement. During the program, youth ages 13-17 years invite their self-identified key adult supports to jointly participate in programming including youth-focused, adult-focused and jointly focused activities. Towards the end of programming participants design and carry out a community project to strengthen intergenerational connections and promote community engagement.
  Arms: Strengthening Connections for Change
Behavioral: Job Readiness Training — Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth.
  Arms: Job Readiness Training

SUMMARY:
This pilot community-partnered cluster-randomized trial will examine the feasibility and acceptability of a social network-based youth violence prevention program called Strengthening Connections for Change for youth ages 13-17 and their key adult supports.

DETAILED DESCRIPTION:
This pilot community-partnered cluster-randomized trial will examine the feasibility and acceptability of a social network-based youth violence prevention program called Strengthening Connections for Change for youth ages 13-17 and their key adult supports. Set in four lower resource Pittsburgh, Pennsylvania neighborhoods, this study brings together youth ages 13-17 and their self-identified key adult supports to focus on leadership, strengthening intergenerational networks, community engagement, and violence prevention.

ELIGIBILITY:
Inclusion Criteria:

Youth:

* Participants must be ages 13-17 (inclusive)
* Participants must speak English

Adults

* Participants must be ages 18 or older
* Participants must speak English

Exclusion Criteria:

Youth:

* Not ages 13-17 (inclusive)
* Do not speak English

Adults

* Less than 18 years of age
* Do not speak English

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants that self report any self-representation of gender identity to include, but not limited to, male, female, trans-male, trans-female, nonbinary, or gender non conforming.
Enrollment: 74 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Culyba, MD PhD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The research team will not make individual participant data (IPD) available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We partnered with youth-serving agencies to assist with recruitment through community settings. During program session #1, youth in the intervention group were asked to identify a key adult support in family, school, or community to participate in the program. The study team reached out to the adult to facilitate enrollment. Of the 34 youth, 11 identified an adult who consented to enroll in the study.
Units Other Than Participants: Neighborhoods
Period: Overall Study
Arm/Group | Strengthening Connections for Change | Job Readiness Training
Started | 45; 2 Neighborhoods (Met eligibility and enrolled in study) | 29; 2 Neighborhoods (Met eligibility and enrolled in study)
Youth Started | 34; 2 Neighborhoods | 29; 2 Neighborhoods
Adults Started | 11; 2 Neighborhoods | 0; 0 Neighborhoods
Youth Completed Baseline Survey | 34; 2 Neighborhoods | 29; 2 Neighborhoods
Adults Completed Baseline Survey | 11; 2 Neighborhoods | 0; 0 Neighborhoods
Youth Completed End of Program Survey | 26; 2 Neighborhoods | 26; 2 Neighborhoods
Adults Completed End of Program Survey | 6; 2 Neighborhoods | 0; 0 Neighborhoods
Completed | 32; 2 Neighborhoods | 26; 2 Neighborhoods
Not Completed | 13; 0 Neighborhoods | 3; 0 Neighborhoods
Not completed — Lost to Follow-up | 13 | 3

BASELINE CHARACTERISTICS:
Population: Two neighborhoods were randomized to the Strengthening Connections for Change (SCC) intervention and two neighborhoods were randomized to Job Readiness Training. In the 2 SCC neighborhoods, both youth and adults were recruited. In the 2 Job Readiness Training neighborhoods only youth were recruited.
Groups:
- Strengthening Connections for Change--Youth: Strengthening Connections for Change uses a group discussion format with activities that explore identity, adolescent-adult relationships, social networks, and community engagement. Youth invite their self-identified key adult supports to jointly participate in programming and curriculum includes youth-focused, adult-focused and jointly focused activities designed to build leadership skills, enhance intergenerational networks, challenge attitudes towards violence and retaliation, and reduce violence involvement. Through 12 sessions (2 hours/session) delivered weekly, Strengthening Connections offers leadership development coupled with strengths-based youth violence prevention programming.
  Strengthening Connections for Change: Strengthening Connections for Change is a 12-session curriculum designed to strengthen adolescent-adult support networks, build leadership skills, foster community engagement, and challenge attitudes and behaviors that foster violence involvement. During the program, youth ages 13-17 years invite their self-identified key adult supports to jointly participate in programming including youth-focused, adult-focused and jointly focused activities. Towards the end of programming participants design and carry out a community project to strengthen intergenerational connections and promote community engagement.
- Strengthening Connections for Change--Adults: During the Strengthening Connections for Change program, youth invite their self-identified key adult supports to jointly participate in programming including youth-focused, adult-focused and jointly focused activities.
- Job Readiness Training--Youth: Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth. Participants receive a 12 session job readiness training with linkages to businesses and employment opportunities. Discussions include a wide range of topics related to career exploration and job readiness.
  Job Readiness Training: Job Readiness Training uses a group discussion format to learn specific skills to prepare for employment including developing goals, seeking jobs, preparing for interviews, and so forth.
- Total: Total of all reporting groups
Arm/Group | Strengthening Connections for Change--Youth | Strengthening Connections for Change--Adults | Job Readiness Training--Youth | Total
Number analyzed (Participants) | 34 | 11 | 29 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8 (1.4) | 47.6 (10.7) | 14.3 (1.4) | 14.6 (1.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-identified gender
  Participants
    Female | 6 | 5 | 16 | 27
    Male | 26 | 5 | 12 | 43
    Non-binary or gender fluid | 0 | 0 | 1 | 1
    Not Reported | 2 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 2 | 8
  Not Hispanic or Latino | 28 | 9 | 27 | 64
  Unknown or Not Reported | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 25 | 8 | 17 | 50
  White | 1 | 0 | 0 | 1
  More than one race | 2 | 1 | 10 | 13
  Unknown or Not Reported | 5 | 2 | 1 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 11 | 29 | 74

OUTCOME MEASURES:

1. Primary Outcome: Participant Attendance
Description: Attendance recorded at beginning and end of each session. Calculated as a proportion of total number of sessions attended (possible session attended #: 0-12 for youth participants and 0-9 for adult participants) using the following method (# youth at session 1 + # youth at session 2 + …)/(# of youth participants x12 sessions) and (# adults at session 1 + # adults at session 2 + …)/(# of adult participants x9 sessions). The possible proportion attended ranges from 0-1.
Time Frame: through intervention completion, 12 weeks
Measure: Number; unit: proportion of sessions attended
Units Other Than Participants: neighborhoods
Groups:
- Strengthening Connections for Change--ADULTS: Strengthening Connections for Change uses a group discussion format with activities that explore identity, adolescent-adult relationships, social networks, and community engagement. Youth invite their self-identified key adult supports to jointly participate in programming and curriculum includes youth-focused, adult-focused and jointly focused activities designed to build leadership skills, enhance intergenerational networks, challenge attitudes towards violence and retaliation, and reduce violence involvement. Through 12 sessions (2 hours/session) delivered weekly, Strengthening Connections offers leadership development coupled with strengths-based youth violence prevention programming.
  Strengthening Connections for Change: Strengthening Connections for Change is a 12-session curriculum designed to strengthen adolescent-adult support networks, build leadership skills, foster community engagement, and challenge attitudes and behaviors that foster violence involvement. During the program, youth ages 13-17 years invite their self-identified key adult supports to jointly participate in programming including youth-focused, adult-focused and jointly focused activities. Towards the end of programming participants design and carry out a community project to strengthen intergenerational connections and promote community engagement.
Arm/Group | Strengthening Connections for Change--YOUTH | Strengthening Connections for Change--ADULTS | Job Readiness Training--YOUTH
Number analyzed (Participants) | 34 | 11 | 29
Number analyzed (neighborhoods) | 2 | 2 | 2
proportion of sessions attended | 0.62 | 0.49 | 0.71

2. Primary Outcome: Participant Overall Satisfaction With Curriculum Content and Format Assessed by Researcher-generated Likert-scale Items
Description: At the end of the program, participants will be asked about how satisfied they were overall with the topics discussed and format of the program using 5-point Likert scale items. Means score will be calculated across the items (possible range: 1-5; higher score means higher satisfaction). This data was collected for the Strengthening Connections for change intervention groups only.
Time Frame: end of program (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: neighborhoods
Arm/Group | Strengthening Connections for Change--YOUTH | Strengthening Connections for Change--ADULTS
Number analyzed (Participants) | 34 | 11
Number analyzed (neighborhoods) | 2 | 2
score on a scale | 3.47 (1.00) | 4.07 (0.70)

3. Secondary Outcome: Participant Satisfaction With Weekly Session Content Assessed by Researcher-generated Likert-scale Items
Description: At the end of each of the 12 sessions, participants will be asked about how satisfied they were with the topics discussed for that session using 5-point Likert scale items. A mean score will be calculated by taking the average of the responses on session forms completed by each youth across all time points (i.e., Session 1 Mean Score + Session 2 Mean Score + Session 3 Mean score +.../ 12 sessions) (possible range: 1-5; higher score means higher satisfaction). This data was collected for the Strengthening Connections for change intervention groups only.
Time Frame: end of program (12 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: neighborhoods
Arm/Group | Strengthening Connections for Change--YOUTH | Strengthening Connections for Change--ADULTS
Number analyzed (Participants) | 34 | 11
Number analyzed (neighborhoods) | 2 | 2
score on a scale | 3.57 (0.96) | 4.32 (0.81)

4. Other Pre Specified Outcome: Change in Social Network Composition
Description: Participants will complete an abbreviated social network survey that asks them to identify key sources of emotional and instrumental support, and to characterize the nature of these relationships (network size, network density, mean link strength).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Violence Perpetration
Description: Summary score of past 30-day youth violence perpetration adapted from the Aggressive Behavior--SAGE Baseline survey (9 items, each measured on a 5-point frequency scale from 0 times to 7 or more times). Violence perpetration items will be added to create a summary violence perpetration score with 1 point for each response of at least 1 time (possible range: 0-9; lower score indicates better outcome).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Change in Violence Victimization
Description: Summary score of past 30-day youth violence victimization adapted from the Victimization--Problem Behavior Frequency Scale (9 items, each measured on a 5-point frequency scale from 0 times to 7 or more times). Violence victimization items will be added to create a summary violence victimization score with 1 point for each response of at least 1 time (possible range: 0-9; lower score indicates better outcome).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Attitudes Towards Violence
Description: Modified from the Children's Perception of Environmental Violence Scale, 6 items assessed on 5-point Likert scale, calculated as a mean score (possible range 1-5; lower score indicates better outcome).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Coping
Description: Modified from the Healthy Pathways Child-Report Scales: Active Coping Scale, 7 items assessed on 5-point Likert scale, calculated as a mean score (possible range 1-5; higher score indicates better outcome).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Future Orientation
Description: Modified from the California Healthy Kids Survey, 7 items assessed on 5-point Likert scale, calculated as a mean score (possible range 1-5; higher score indicates better outcome).
Time Frame: Baseline, end of program (12 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was recorded for the duration of their involvement as a research participant. Data was collected across the full study from enrollment of the first participant to study completion (up to 12 weeks).
Description: We follow the definitions of adverse events as outlined by the clinicaltrials.gov definitions and University of Pittsburgh Human Subjects Research Protection Office, and any questions we have about specific events, we review with a representative from this office.
Arm/Group | Strengthening Connections for Change--YOUTH | Strengthening Connections for Change--ADULTS | Job Readiness Training
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/11 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/11 | 0/29
Other Adverse Events (participants affected / at risk) | 0/34 | 0/11 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT05185453/Prot_SAP_000.pdf